CLINICAL TRIAL: NCT01799135
Title: Feasibility Study of the Utility of Pulmonary Dynamic Contrast Enhanced MRI for Assessment of Tumor Response and Lung Injury and for Treatment Planning for Stereotactic Body Radiation Therapy for Early Stage Non-Small Cell Lung Cancer
Brief Title: Feasibility Study of Enhanced MRI for Early Stage Non Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Raymond H. Mak, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-004
Record Dates: First submitted 2012-12-11; First posted 2013-02-26 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Arm (Experimental): Stereotactic Body Radiation Therapy: either 54 Gy in 3 fractions or 50-60 Gy in 5 fraction over a span of 15 days at most.
  DCE-MRI was performed at four time points during therapy: at baseline prior to SBRT, 1-2 days after the first treatment fraction, 1-2 weeks after the end of the SBRT course, and 3 months after completing radiotherapy.
  4D-CT scan 3 months after completing radiotherapy.
  Interventions: Other: DCE-MRI scan; Radiation: Stereotactic Body Radiation Therapy; Other: 4D-CT scan

INTERVENTIONS:
Other: DCE-MRI scan
Radiation: Stereotactic Body Radiation Therapy
Other: 4D-CT scan

SUMMARY:
This is a pilot study. A pilot study is done with a small number of participants to see if a technique works before using it in a larger research study. This pilot study is evaluating a special kind of MRI scan of the lungs called dynamic contrast enhanced MRI (DCE-MRI).

DCE-MRI can demonstrate how much blood flows through the tumor and lungs and tell us how active the tumor is, as well as how functional the lungs are. As part of this scan, participants will receive an intravenous (into the blood via puncture of a vein) injection of gadolinium contrast, a dye that helps us see the tumor and lung tissue more clearly. Gadolinium is approved by the FDA and is routinely used for MRI.

The goal of the study is to determine whether DCE-MRI can provide images of the response of the tumor and the normal lung tissue to SBRT and to potentially hep improve treatment-planning methods for patients treated with SBRT in the future. We will also study how the final DCE-MRI scan compares with another form of imaging, called 4-dimensional computed tomography (4D-CT), that looks at the breathing capacity of the lungs. Although we are researching the usefulness of DCE-MRI in early stage non-small cell lung cancer treated with SBRT in this study, DCE-MRI with the dye injection is not an experimental technology and is routinely used in the clinic for other indications. The 4D-CT scan is also not experimental and is used for radiation planning and imaging of the lungs.

The SBRT you will receive will be standard treatment and will not be affected by your participation in this study or by these DCE-MRI scans. That means that the findings on the scan will not be used to alter your planned treatment in any way. Additionally, participants will undergo the routine work-up prior to SBRT and surveillance studies after treatment is complete.

DETAILED DESCRIPTION:
If you agree to participate in this research study you will be asked to undergo some screening tests or procedures to find out if you can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history, performance status, physical exam, assessment of tumor, assessment of breathing function and blood tests. We will also confirm that you have no contraindications to MRIs. If these tests confirm that you are eligible to participate in the research study, you will begin the study scans. If you do not meet the eligibility criteria you will not be able to participate in this research study.

If you qualify for this research study, you will come for the first study visit that will last about one and a half hours. We will use the first 30 minutes to make sure you can undergo a MRI scan (MRI screening).

Before the MRI scan, we will explain how we want you to breathe during the scan. You will breathe in small and regular breaths for one part of the exam. In another part of the exam, you will hold your breath as much as possible and breathe in between breath-holds.

An MRI contrast agent called gadolinium will be injected into a vein in your arm through an intravenous (IV) line. A contrast agent is a dye that is injected into the body to allow for better visualization (images) during an MRI exam.

You will be aked to lie down on your back on a platform that can slide into the scanner. The scan will last 60 minutes. You will hear a loud knocking or hammering noise while the MRI is taking pictures, but the process itself will be painless. You will be given disposable earplugs to help make the noise less noticeable.

During the procedure, you will be able to talk to the MRI technician through an intercom. If you feel too uncomfortable to continue the scan for any reason, the procedure will be immediately stopped and you will be removed from the MRI scanner.

You will then undergo a standard treatment planning session for SBRT. This will include a standard 4D-CT scan and a standard planning CT scan. As part of the standard planning CT scan, an intravenous (IV, through a vein) line will be placed, and you will receive an injection of IV contrast. The planning process will be conducted exactly as it would if you were not participating in this research study; it is not experimental in any way.

One to two weeks later, you will start standard SBRT treatment for your early stage non-small cell lung cancer. This treatment will be delivered exactly as it would if you were not participating in this research study; it is not experimental in any way.

After the first treatment, you will undergo your second study DCE-MRI, which is identical to the initial DCE-MRI scan as described above.

You will then have two more study visits for the post-treatment research scans. The first visit will occur 1-2 weeks after completion of SBRT. It will involve a 30-minute routine clinic visit with your radiation oncologist to assess your recovery from treatment, and then you will undergo your third study DCE-MRI, which is identical to the DCE-MRI scans described above.

You will then undergo the fourth (final) study DCE-MRI scan 3-4 months after completion of SBRT. This scan will be identical to the three previous DCE-MRI scans. At this visit, you will also have a repeat 4D-CT scan which is study related. You will also have a routine clinic visit with your radiation oncologist at this time. You will then undergo the standard post-treatment re-evaluation imaging including a repeat PET/CT and a pulmonary function test.

Once you have completed the DCE-MRI scans, no further study follow-up will be necessary. However, you will continue with routine follow-up with your radiation oncologist as part of standard care. You will be in this research study for approximately four months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* Tumor between 1 cm and 6 cm
* No evidence of nodal involvement or distant metastases
* Deemed to be a candidate for stereotactic body radiation therapy for NSCLC
* Able to lie still during DCE-MRI (up to 60 minutes)
* Adequate renal function to tolerate intravenous gadolinium contrast injection

Exclusion Criteria:

* Prior thoracic radiotherapy or surgery
* Implanted pacemaker or cardiac defibrillator
* Contraindications to undergoing MRI
* Uncontrolled intercurrent illness
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-11; Primary Completion 2019-01 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Mak, MD, Principal Investigator — Dana-Farer Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 2012 to August 2016
Groups:
- Experimental Arm: Stereotactic Body Radiation Therapy: either 54 Gy in 3 fractions or 50-60 Gy in 5 fraction over a span of 15 days at most.
  DCE-MRI was performed at four time points during therapy: at baseline prior to SBRT, 1-2 days after the first treatment fraction, 1-2 weeks after the end of the SBRT course, and 3 months after completing radiotherapy.
  4D-CT scan 3 months after completing radiotherapy.
  DCE-MRI scan
  Stereotactic Body Radiation Therapy
  4D-CT scan
Period: Overall Study
Arm/Group | Experimental Arm
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: year] | 67.5 [59 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Rate at 1-2 Days After the First SBRT Treatment and 1-2 Weeks and 3-4 Months After SBRT Treatment.
Description: Feasibility rate is defined as the number of participants with a 20% or greater change in tumor perfusion at 1-2 days, 1-2 weeks, and 3-4 months from baseline. Feasibility must be achieved at all 3 timepoints to be considered as a success.
  Perfusion measured using establish methods in conjunction with Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI)
Time Frame: Measured 1-2 days, 1-2 weeks, and 3-4 months from baseline.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
percentage of participants | 66.7 [27.1 to 93.7]

2. Secondary Outcome: Feasibility Rate of Using Pulmonary DCE-MRI in Characterizing Acute and Subacute Radiation-induced Lung Injury
Description: Feasibility (success) is defined as successfully enrolling patients, processing the pulmonary DCE-MRI data, and observing at least a 20% change in perfusion on the 3-month scan.
Time Frame: 3 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
percentage of participants | 50 [15.3 to 84.6]

3. Secondary Outcome: Feasibility Rate of Using 4D-CT Ventilation Imaging With Pulmonary DCE-MRI in Characterizing Acute and Subacute Radiation Induced Lung Injury
Description: Feasibility (success) is defined as successfully enrolling patients, processing the pulmonary DCE-MRI and 4D-CT data, and observing at least a 20% change in perfusion on the 3-month scan.
Time Frame: 3 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
percentage of participants | 0 [0 to 39.3]

4. Secondary Outcome: Feasibility Rate of Using Pulmonary DCE-MRI to Identify Regions of Functional Lung for SBRT Treatment Planning
Description: Feasibility will be defined as the ability to perform a retrospective comparative treatment planning study using the DCE-MRI images acquired prior to treatment for each participant. Regions of functional and non-functional lung will be defined on each MRI, and the images will be registered to the 4DCT used for treatment planning. The functional-lung contours will be transferred to the 4D-CT based on this registration. the treatment plan will attempt to maximize sparing of functional-lung regions while maintaining adequate target coverage and not exceeding other normal-tissue constraints. The functional-lung based treatment plans generated in this manner will be compared to the corresponding standard plans that were used to treat the patient. Changes in the functional-lung V20 and V5 will be used to analyze changes in functional-lung sparing
Time Frame: 3 months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Experimental Arm
Number analyzed (Participants) | 6
percentage of participants | 83.3 [41.8 to 99.1]

ADVERSE EVENTS:
Time Frame: Up to 4 months
Description: Serious Adverse Events (SAE's) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term
Arm/Group | Experimental Arm
All-Cause Mortality (participants affected / at risk) | 1/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental Arm (N=6)
Death NOS (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Arm (N=6)
Hypertension (Vascular disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-28): https://cdn.clinicaltrials.gov/large-docs/35/NCT01799135/Prot_SAP_000.pdf